CLINICAL TRIAL: NCT01674179
Title: Quantitative EEG During PSG in Patients With and Without Fibromyalgia
Acronym: FMQEEG-10-26
Status: Completed | Type: Observational
Sponsor: SouthCoast Medical Group (Other)
Responsible Party: Principal Investigator, Victor Rosenfeld MD, Principal Investigator, SouthCoast Medical Group
Other Study IDs: SM 10-26
Record Dates: First submitted 2010-09-10; First posted 2012-08-28 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; qEEG; Sleep; Pain
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ACR diagnosis of Fibromyalgia
- Patients without Fibromyalgia

SUMMARY:
The purpose of this study is to retrospectively analyze Clinical and Nocturnal Polysomnographic Data (Overnight Sleep Studies) in patients with and without Fibromyalgia.

Fibromyalgia is a pain syndrome associated with dysfunctional sleep, fatigue, frequent awakenings, non-refreshing sleep, and alpha frequency intrusions. Quantitative EEG during routine Nocturnal Polysomnography can be used to assess Alpha/Delta sleep. Hypothesis: Alpha intrusions may be an objective marker for Fibromyalgia and may correlate with current clinical American College of Rheumatology Criteria for the diagnosis of Fibromyalgia.

DETAILED DESCRIPTION:
This is a Retrospective Study of patients with and without Fibromyalgia seen in private practice from Aug 2007-July 2010 who underwent Overnight Sleep Studies (PSG)

The polysomnographic and clinical data from research subjects with a diagnosis of Fibromyalgia will be compared to other subjects' PSG and Clinical data who were also referred for Sleep Studies including those with Sleep Apnea, Narcolepsy, Periodic Limb Movement, Fatigue, and Insomnia which are standard indications for Overnight Sleep Studies.

Clinical Data: Clinical Data points will include the following: 1. Research Study Number, 2. Age, 3. Gender, 4. Body Mass Index, 5. Epworth Sleepiness Scale (self reported scale on Sleepiness), 6. Fatigue Severity Scale (self reported scale on Fatigue, 7. American College of Rheumatology (ACR) Criteria for Fibromyalgia, 8. Manual Tender Point Exam (# of anatomically specific tender points/18), 9. Medications: Benzodiazepines (Bnz, Bnz ), Tricyclic Antidepressants (TCA) and Serotonin Reuptake Inhibitors (SSRIs SNRIs).

Sleep Study Data Points: The following data points will be captured from Overnight Sleep Studies: 1. Total Sleep Time, 2. Sleep Efficiency, 3. Wake After Sleep Onset, 4.Apnea/Hypopnea Index, 5. Respiratory Distress Index, 6. Periodic Limb Movement Index, 7. Periodic Limb Movement Arousal Index, and 8. Quantitative EEG: Delta Event/Alpha Event Ratio.

ELIGIBILITY:
Inclusion Criteria:

* Completed a polysomnogram
* Complaints of disordered sleep
* Age 18 to 80 inclusive
* Men and women

Exclusion Criteria:

* History of seizure
* use of benzodiazepines
* use of AEDs
* any significant medical condition other than disorder sleep or fibromyalgia that would influence qEEG measures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Private Sleep Practice
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Delta Event/Alpha Event Ratios in Non-REM sleep | up to 24 weeks
  Assess the sensitivity and specificity of Delta Event/Alpha Event Ratios in Non-REM sleep in patients with and without Fibromyalgia

CONTACTS AND LOCATIONS:
Overall Officials: Victor Rosenfeld, MD, Principal Investigator — SouthCoast Medical Group
Locations (1):
- SouthCoast Medical Group, Savannah, Georgia, United States

REFERENCES:
- [Derived] Rosenfeld VW, Rutledge DN, Stern JM. Polysomnography with quantitative EEG in patients with and without fibromyalgia. J Clin Neurophysiol. 2015 Apr;32(2):164-70. doi: 10.1097/WNP.0000000000000134. PMID 25233248